CLINICAL TRIAL: NCT05010421
Title: CO2 Non-ablative Laser Versus Topical Clobetasol for Lichen Sclerosus: a Prospective, Open-label, Randomized Trial
Brief Title: Laser vs Clobetasol for Lichen Sclerosus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LASER-LICH1
Record Dates: First submitted 2021-07-16; First posted 2021-08-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lichen Sclerosus
Keywords: Lichen Sclerosus; Laser; Clobetasol; Corticosteroids
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus | interventions — Clobetasol

STUDY DESIGN:
Intervention Model Description: Prospective randomized open single center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clobetasol Group (Active Comparator): Treatment with clobetasol-0,05% over 3 months (month 1: daily, month 2: every other day, month 3: 3x per week)
  Interventions: Drug: Clobetasol 0.05% Emollient Top Cream
- Laser Group (Experimental): 3 applications every 14 days of a non-ablative CO2 laser treatment
  Interventions: Device: Non-ablative CO2 Laser

INTERVENTIONS:
Drug: Clobetasol 0.05% Emollient Top Cream — Topical corticosteroid treatment of affected vulvar skin areas.
  Other Names: Dermoxin (Germany), Temovate, Clobex, Dermovate, Impoyz
  Arms: Clobetasol Group
Device: Non-ablative CO2 Laser — Superficial non-ablative laser treatment of affected vulvar skin areas.
  Arms: Laser Group

SUMMARY:
Lichen sclerosus (LS) is a common autoimmune disease of the genital skin. It affects 1/900 women with an age peak in the sixth decade of life and is manifested by chronic inflammation of the genital, perineal, and perianal areas associated with itching, burning, pain, and soreness. In addition, LS is associated with an increased risk of vulvar cancer.

Treatment options for LS include topical steroids such as clobetasol, immunomodulators such as tacrolimus, and non-ablative laser treatment. Although both treatments are well documented and used in clinical practice, direct comparative studies of the efficacy of topical corticosteroids versus laser treatment in women with LS are rare. For example, a PubMed literature search (search date 2021-03-14; search terms: lichen sclerosus, laser, corticosteroids, steroids, clobetasol, randomized) identified only a single randomized trial with limited power.

Given the available evidence, further high-quality studies are needed to define the superiority/inferiority of the different available treatment options such as nonablative lasers and topical corticosteroids.

Therefore, in this prospective, randomized, open-label, comparative study, treatment success after 3 courses of non-ablative treatment with CO2 laser every 14 days will be compared with treatment success after topical application of clobetasol 0.05% over 3 months (daily in the first month, every other day in month 2, and 3 times/week during month 3) at the time point 3 months after treatment initiation.

DETAILED DESCRIPTION:
Lichen sclerosus (LS) is a common autoimmune disorder of the genital skin. It affects 1/900 women with an age peak in the sixth decade of life. LS is a chronic inflammatory condition affecting the genital, perineal, and perianal areas and causes itching, burning, pain, and soreness. Histologically, LS is characterized by epidermal atrophy, hyperkeratosis, follicular plugging, degeneration of the basal layer, and subepidermal hyalinization of collagen in the papillary dermis with a lymphocytic infiltrate. Affected women typically suffer significant long-term genital damage including scarring, fusion of the vulval labia, narrowing of the vaginal opening, dyspareunia, and burying of the clitoris. In addition, LS is associated with an increased risk of vulvar cancer.

Treatment options of LS include topical steroids such as clobetasol, topical immunomodulators such as tacrolimus, and non-ablative laser treatment. In a systematic review of the literature with 7 studies and 249 participants, clobetasol achieved improvement rates and remission rates of 70% to 89% and 20% to 35%, respectively. In comparison, non-ablative laser treatment leads to significant improvements in vulvar itching, dryness, pain, and dyspareunia in 50% to 85% of women with remission rates of up to 80% after 14 years of follow-up. Although both treatments are well documented and used in clinical practice, direct comparative studies assessing the efficacy of topical corticosteroids versus laser treatment in women with LS are rare. For example, in a PubMed literature search (search date 2021-03-14; search terms: lichen sclerosus, laser, corticosteroids, steroids, clobetasol, randomized) only one randomized trial was identified. In this study, the authors included 40 women with LS and compared 3 applications of non-ablative laser 2 weeks apart with 4 weeks of twice daily (2 weeks), once daily (1 week), and every other day (1 week) of topical clobetasol 0.05% cream. After 3 months of treatment laser-treated women had a significantly higher sum score (including burning, itching, and pain) measured on an 11-step visual analogue scale (VAS). Both treatments demonstrated histological improvement with reductions of inflammatory hallmarks in skin biopsies.

Given this body of evidence, more high-quality studies are needed to define the superiority/inferiority of the different available treatment options such as non-ablative laser and topical corticosteroids. Therefore, a prospective, randomized trial comparing non-ablative CO2 laser treatment and topical clobetasol 0.05% will be conducted. The aim of this prospective, randomized, open-label, comparative trial is to establish or refute the superiority of 3 courses of non-ablative treatment by CO2 laser every 14 days compared to topical clobetasol 0.05% (daily in month 1, every other day in month 2, and 3 times/week in month 3) for 3 months. The primary endpoint of this study is a sum score including the pathognomonic symptoms of LS, namely vulvar burning, itching, and pain, each measured on an 11-step VAS. Secondary endpoints will include the physician-scored rate of visual improvement (measured on an 11-item VAS), side effects, and patient-reported outcomes such as subjective overall improvement, general satisfaction, and quality of life (measured by a validated questionnaire for vulval disorders; i.e. the VDQI (Vulval Disease Quality of Life Index).

ELIGIBILITY:
Inclusion Criteria:

* Women, age ≥ 18 years
* Established diagnosis of LS (vulva and/or perineum and/or perianal region)
* Willingness to comply with study requirements
* No significant language barrier

Exclusion Criteria:

* Concurrent immunosuppressive treatment
* A history of vulvar cancer and/or vulvar dysplasia
* A history of vulvar surgery
* A contraindication against clobetasol treatment
* A known sun light allergy
* A known skin condition interfering with local ablative treatment such as neurodermatitis or bullous pemphigoid

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Vulvar burning, itching, and pain | from date of randomization until 12 weeks
  Summary score of three symptoms of LS, i.e. vulvar burning, itching, and pain (11-item VAS each).
  Higher values mean worse outcome.

SECONDARY OUTCOMES:
Efficacy - Physician-scored rate of visual improvement (0-10) | 3 months after treatment start
  11-item VAS; higher values mean better outcome.
Safety - Number and severity of side effects | 0-7 days after laser treatment (laser group); as well as throughout study duration (3 months; both groups)
  Side effects (perioperative and postoperative complications up to 7 days) including but not limited to bleeding, infection, wound breakdown, unscheduled re-admission, and local pain necessitating systemic analgesia.
Subjective overall improvement (0-10) | 3 months after treatment start
  The patient's subjective judgement of improvement (11-item VAS); higher values mean better outcome.
Vulval Disease Quality of life Index (0-45) | Throughout study completion (3 months; for a total of 4 or 5 assessments, depending on group assignment)
  Quality of life assessed before the start of therapy, after every treatment course (laser group; days 0, 14, 28, 42) or after 2 and 6 weeks (clobetasol group; days 0, 14, 42), and after 3 months (both groups) using a standardized, validated questionnaire (VDQI, Vulval Disease Quality of life Index). Lower score mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, Principal Investigator — Ruhr-Universität Bochum / Marien Hospital Herne
Locations (1):
- Marien Hospital Herne, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request made to the corresponding author. This includes individual participant data underlying the results presented here, after deidentification, as well as data dictionaries and the the study protocol. Data is available after publication, without a specific end date. Requesting investigators must show that their proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication of the study results, no time limit.
Access Criteria: Reasonable request, approval of the intended study by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Bizjak Ogrinc U, Sencar S, Luzar B, Lukanovic A. Efficacy of Non-ablative Laser Therapy for Lichen Sclerosus: A Randomized Controlled Trial. J Obstet Gynaecol Can. 2019 Dec;41(12):1717-1725. doi: 10.1016/j.jogc.2019.01.023. Epub 2019 Apr 11. PMID 30981618
- [Background] Felmingham C, Chan L, Doyle LW, Veysey E. The Vulval Disease Quality of Life Index in women with vulval lichen sclerosus correlates with clinician and symptom scores. Australas J Dermatol. 2020 May;61(2):110-118. doi: 10.1111/ajd.13197. Epub 2019 Nov 14. PMID 31729009
- [Background] Murphy R. Lichen sclerosus. Dermatol Clin. 2010 Oct;28(4):707-15. doi: 10.1016/j.det.2010.07.006. PMID 20883914
- [Background] Renaud-Vilmer C, Cavelier-Balloy B, Porcher R, Dubertret L. Vulvar lichen sclerosus: effect of long-term topical application of a potent steroid on the course of the disease. Arch Dermatol. 2004 Jun;140(6):709-12. doi: 10.1001/archderm.140.6.709. PMID 15210462
- [Background] Chi CC, Kirtschig G, Baldo M, Lewis F, Wang SH, Wojnarowska F. Systematic review and meta-analysis of randomized controlled trials on topical interventions for genital lichen sclerosus. J Am Acad Dermatol. 2012 Aug;67(2):305-12. doi: 10.1016/j.jaad.2012.02.044. Epub 2012 Apr 6. PMID 22483994
- [Background] Pagano T, Conforti A, Buonfantino C, Schettini F, Vallone R, Gallo A, Avino L, Alviggi C, De Placido G, Sopracordevole F. Effect of rescue fractional microablative CO2 laser on symptoms and sexual dysfunction in women affected by vulvar lichen sclerosus resistant to long-term use of topic corticosteroid: a prospective longitudinal study. Menopause. 2020 Apr;27(4):418-422. doi: 10.1097/GME.0000000000001482. PMID 31934950